CLINICAL TRIAL: NCT07405489
Title: A Retrospective Comparative Cohort Study Evaluating the Efficacy, Anatomical Outcomes, Recurrence Rates, and Safety of Oral Prednisolone Versus Posterior Sub-Tenon Triamcinolone Acetonide as Initial Therapy in Acute Ocular Vogt-Koyanagi-Harada Disease
Brief Title: Oral Prednisolone Versus Posterior Sub-Tenon Triamcinolone for Acute Ocular VKH
Acronym: VKH-OC
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Collaborators: faculty of medicine, Benha university (Unknown)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Other Study IDs: VKH Treatment; Benha University (Other: Al-Azhar University)
Record Dates: First submitted 2026-01-30; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: VKH Syndrome
Keywords: Vogt-Koyanagi-Harada disease; acute uveitis; optical coherence tomography
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Prednisolone Group: Patients received oral prednisolone at 1 mg/kg/day (maximum 80 mg/day) as initial therapy for acute ocular VKH. The full dose was given for ~1 week followed by gradual taper over 3-6 weeks. Topical corticosteroids and cycloplegics were allowed as adjunct therapy.
- Posterior Sub-Tenon Triamcinolone (PST/STA) Group: Patients received a posterior sub-Tenon injection of triamcinolone acetonide (40 mg/1 mL) as initial therapy for acute ocular VKH. A second injection at 4-6 weeks was administered if residual inflammation persisted. Systemic steroids were not used unless rescue criteria were met.

SUMMARY:
Vogt-Koyanagi-Harada (VKH) disease is a rare autoimmune disorder characterized by bilateral ocular inflammation that may lead to serous retinal detachment and permanent visual impairment if not promptly treated. Systemic corticosteroids are commonly used as first-line therapy; however, periocular corticosteroid administration has been proposed as an alternative approach that may reduce systemic adverse effects.

This retrospective cohort study reviewed the medical records of patients with acute ocular VKH disease to compare two initial treatment strategies: systemic oral prednisolone and posterior sub-Tenon triamcinolone acetonide (PST/STA). The primary objective was to evaluate control of ocular inflammation three months after treatment initiation. Secondary objectives included assessment of visual acuity changes over six months, anatomical recovery on optical coherence tomography (OCT), recurrence of inflammation, need for additional therapy, and treatment-related adverse events.

DETAILED DESCRIPTION:
This retrospective comparative observational cohort study evaluated the efficacy and safety of oral prednisolone versus posterior sub-Tenon triamcinolone acetonide (PST/STA) as initial therapy for acute ocular Vogt-Koyanagi-Harada (VKH) disease. The study was conducted at the Ophthalmology Department, Faculty of Medicine, Benha University, Egypt, through a review of electronic and paper-based medical records of patients treated between January 2021 and December 2025.

Eligible patients were adults diagnosed with acute ocular VKH disease who had not received prior systemic or periocular corticosteroid therapy and who had a minimum follow-up duration of six months. Patients were managed according to routine clinical practice and received either systemic oral prednisolone or PST/STA as initial treatment, based on treating physician discretion. Both eyes of each patient were treated using the same modality, and analyses were performed at the patient level.

Patients in the oral prednisolone group received an initial dose of approximately 1 mg/kg/day (maximum 80 mg/day), followed by gradual tapering over 3-6 weeks. Patients in the PST/STA group received a posterior sub-Tenon injection of triamcinolone acetonide (40 mg/1 mL), with repeat injection considered if clinically indicated. Topical corticosteroids and cycloplegics were permitted in both groups. Systemic corticosteroids were reserved as rescue therapy in the PST/STA group when necessary.

Data extracted from medical records included demographic characteristics, baseline ophthalmic findings, best-corrected visual acuity (BCVA), OCT parameters, follow-up clinical assessments, recurrence episodes, requirement for rescue therapy, and ocular or systemic adverse events. The primary outcome measure was control of ocular inflammation at three months following initiation of therapy. Secondary outcome measures included longitudinal changes in BCVA, OCT-based anatomical recovery, recurrence of inflammation, need for additional treatment, and treatment-related adverse events during follow-up.

Statistical analysis was planned using appropriate parametric or non-parametric tests for between-group comparisons, survival analysis methods for time-to-event outcomes, and a significance threshold of p < 0.05.

The study protocol was approved by the Institutional Review Board of the Faculty of Medicine, Benha University (Approval No. RC 11_1_2026). Due to the retrospective nature of the study, informed consent was waived. The study was conducted in accordance with the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

Diagnosis of definite or probable acute ocular Vogt-Koyanagi-Harada (VKH) disease

Active intraocular inflammation (choroiditis, serous retinal detachment, or panuveitis)

No prior treatment for the current VKH episode

Minimum follow-up of 6 months with complete medical records, including BCVA and OCT data

Exclusion Criteria:

* Prior systemic or periocular corticosteroid therapy for VKH

Use of immunosuppressive or biologic agents at presentation

Pre-existing glaucoma, ocular hypertension, or advanced cataract

Retinal diseases affecting visual outcomes (e.g., diabetic retinopathy, age-related macular degeneration)

Incomplete medical records or missing OCT/BCVA data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included treatment-naïve adult patients with acute ocular VKH disease who received either oral prednisolone or posterior sub-Tenon triamcinolone acetonide as initial therapy. All patients had bilateral disease; both eyes received the same treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Complete Control of Ocular Inflammation at 3 Months | 3 months from treatment initiation
  Complete control of ocular inflammation is defined as a composite outcome, achieved when all of the following criteria are met at the 3-month visit:
  Absence of active intraocular inflammation on clinical examination
  Complete resolution of subretinal fluid on optical coherence tomography (OCT)
  Stable or improved best-corrected visual acuity (BCVA) compared with baseline
  Unit of Measure: Proportion of participants (%)

SECONDARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) | Baseline, 1 month, 3 months, and 6 months
  Change in BCVA measured in logarithm of the minimum angle of resolution (logMAR) units during follow-up.
Resolution of Subretinal Fluid on Optical Coherence Tomography (OCT) | Baseline, 3 months, 6 months
  Presence or absence of subretinal fluid on OCT imaging during follow-up.
Change in Central Macular Thickness (CMT) | Baseline, 3 months, and 6 months
  Change in central macular thickness measured by OCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Benha, Egypt